CLINICAL TRIAL: NCT01102725
Title: The Challenge of Assessing Infectious Risk and Visceral Closure in NOTES: A Prospective Study Examining Routine Colorectal Surgery as a Model in Humans
Brief Title: Assessing Infectious Risk and Visceral Closure in Natural Orifice Translumenal Endoscopic Surgery (NOTES)
Acronym: NOTES
Status: Completed | Type: Observational
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Jeffrey Marks, MD, Director, Surgical Endoscopy, University Hospitals Cleveland Medical Center
Other Study IDs: 02-09-39; 02-09-39 (Other: University Hospital Case Medical Center)
Record Dates: First submitted 2010-04-12; First posted 2010-04-13 (Estimated); Last update posted 2014-12-16 (Estimated); Status verified 2014-12

CONDITIONS: Colonic Diseases; Rectal Diseases
Keywords: Colon Surgery; Rectal Surgery; Colorectal Surgery
MeSH Terms: conditions — Colonic Diseases; Rectal Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Colorectal Surgery: Subject who are undergoing a colon or rectal resection

SUMMARY:
The purpose of this study is to determine:

1. What quantity of bacteria is spilled into the abdomen during a colon resection
2. If there is a correlation between the quantity and post-operative infection
3. What intralumenal pressure is generated when testing the colonic anastomosis for air leak

DETAILED DESCRIPTION:
The acceptance and advancement of natural orifice translumenal endoscopic surgery (NOTES) has forced investigators to challenge many firmly accepted surgical practices. The most obvious one being: violating a remote hollow viscous that is uninvolved in the desired surgical intervention. This of course brings into question (1) "How much peritoneal contamination can be tolerated without raising infection risk?" and (2) "How will one repair this intended visceral injury?" This study is intended to bring to light what has been done in animal models, and further, how it will translate in to the now more important human arena.

In this study, patients who are undergoing an elective colectomy will be investigated to quantify what amount of peritoneal contamination is tolerated despite rare abscess formation occurring. Subject will undergo peritoneal washings before and after colonic resection to measure the bacterial load spilled. This data would be beneficial to support that patients who are undergoing a NOTES procedure can and will be able to tolerate a definite quantity of bacterial contaminate. Furthermore, by observing the exact values of peritoneal contamination present there may be a certain level to which infectious complication are more likely to occur. This may provide some insight in NOTES as to when patients may benefit post-operatively from a prophylactic course of antibiotic therapy in response to their higher than tolerable intra-peritoneal bacterial load.

The other component to this study will be to challenge how investigators are examining closure devices in the animal model. Many researchers, including authors of this protocol, have utilized bursting pressure as an objective test to assess the integrity of a completed closure. Current surgical practice uses the insufflation of an endoscope or even a bulb syringe to test for leak of a colonic anastomosis. We intend to measure the pressures that are achieved in a clinical setting to determine the bursting pressures that are required to assess NOTES closure and eliminate the likely unsupported value being placed on a higher bursting pressure commonly quoted in NOTES closure studies.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female patients ≥18 years of age
* Subjects have a known preexisting condition that has been deemed treatable by totally laparoscopic or hand-assisted laparoscopic colorectal resection
* Any colon or rectal resection where ileocolonic, ileorectal, colocolonic, or colorectal anastomoses is created in the pelvis requiring a leak test. Air-leak test can be performed by an instrument of the surgeons discretion, such as a colonoscope, sigmoidoscope (rigid or flexible), or bulb syringe.

Exclusion Criteria:

* Surgical resection performed in an emergency setting
* Patients undergoing resection in a known contaminated field (i.e. entero-/colo-cutaneous fistula or acute diverticulitis) as this will bias the bacterial cultures collected intraoperatively

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Our institution performed over 200 laparoscopic colon resections in the past year and should have no trouble accruing the number of patients required for the study. Subjects will be recruited until 90 patients have been enrolled. We will not specifically recruit or specifically exclude potential patients on the basis of their race or on the basis of our study demographics to date. No vulnerable subjects will be recruited into this study as this study will prolong the surgery by approximately 15 minutes which can be significant in the vulnerable population such as pregnant women and minors. Potential subjects who meet inclusion criteria will be approached for possible participation during a pre-operative clinic visit or on the day of surgery in the pre-operative area.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2010-04; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey M. Marks, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Case Medical Center, Cleveland, Ohio, United States